CLINICAL TRIAL: NCT00554619
Title: Study AMB107818, Clinical Evaluation of GSK1325760A in the Treatment of Pulmonary Arterial Hypertension (PAH)- An Open Label Study of GSK1325760A to Evaluate the Safety and Efficacy of GSK1325760A - a Long-term Extension Study -
Brief Title: A Study to Evaluate GSK1325760A - a Long-Term Extension Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMB107818
Record Dates: First submitted 2007-11-05; First posted 2007-11-07 (Estimated); Results first posted 2012-02-13 (Estimated); Last update posted 2012-11-05 (Estimated); Status verified 2012-10

CONDITIONS: Pulmonary Arterial Hypertension; Hypertension, Pulmonary
Keywords: Pulmonary Arterial Hypertension; Ambrisentan
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Hypertension, Pulmonary | interventions — ambrisentan

ARMS (1):
- GSK1325760A (Experimental)
  Interventions: Drug: GSK1325760A

INTERVENTIONS:
Drug: GSK1325760A — 2.5mg, 5mg or 10mg/day, po, GSK1325760A treatment will be continued until its approval by the MHLW.

SUMMARY:
The primary objective of this study is to evaluate the safety of long-term administration of GSK1325760A in patients with PAH.

The secondary objectives of this study are to evaluate long-term administration of GSK1325760A on:

* Improvement in exercise capacity (six-minutes walk distance: 6MWD), change in WHO Functional Classification and time to clinical worsening of PAH
* Change in the Borg Dyspnea Index (assessed immediately following the six-minute walk test [6MWT])
* Change in plasma brain natriuretic peptide (BNP) levels
* Cardiopulmonary hemodynamics parameters (as measured by echocardiography)

ELIGIBILITY:
Inclusion Criteria:

* Subjects who complete the 24-week administration of the Phase II/III study (Study No.AMB107816)
* Subjects who are assessed that the long-term extension administration of GSK1325760A is appropriate in the judgement of the investigator or subinvestigator
* Subjects who request the long-term extension administration of GSK1325760A, and agree to newly sign the informed consent form

Exclusion Criteria:

* Subjects who have been withdrawn from the Phase II/III study.
* Female subjects who wish to become pregnant.
* Treatment with other PAH medication is needed.
* A worsening of 2 or more levels of the WHO Functional Classification (see Appendix 2.1) comparing with the baseline of Phase II/III study (Study No.AMB107816).
* Worsening of right ventricular failure (e.g. as indicated by increased jugular venous pressure, new/worsened hepatomegaly, ascites, or peripheral edema) during Phase II/III study (Study No.AMB107816).
* Rapidly progressing cardiac, hepatic or renal failure during Phase II/III study (Study No.AMB107816).
* Participation to the long-term extension study is considered as inappropriate in the judgment of the investigator or subinvestigator.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2008-02; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (9):
- Japan (9):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Ishikawa
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Kyoto
  - GSK Investigational Site, Okayama
  - GSK Investigational Site, Okinawa
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Tokyo

REFERENCES:
- [Derived] Yoshida S, Shirato K, Shimamura R, Iwase T, Aoyagi N, Nakajima H. Long-term safety and efficacy of ambrisentan in Japanese adults with pulmonary arterial hypertension. Curr Med Res Opin. 2012 Jun;28(6):1069-76. doi: 10.1185/03007995.2012.685930. Epub 2012 May 15. PMID 22506623

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study AMB107818 was an extension study of Study AMB107816 (NCT00540436).
Groups:
- GSK1325760A: Dose of GSK1325760A could be adjusted up to 10 milligrams, once daily, as appropriate according to a participant's condition.
Period: Overall Study
Arm/Group | GSK1325760A
Started | 21
Completed | 18
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — Physician Decision | 1
Not completed — Liver Function Test Abnormality | 1

BASELINE CHARACTERISTICS:
Arm/Group | GSK1325760A
Number analyzed (Participants) | 21
Age Continuous [Mean (Standard Deviation); unit: Years] | 45.6 (12.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 3
Race/Ethnicity, Customized [Number; unit: participants]
  Asian - Japanese Heritage | 21

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Adverse Event
Description: An adverse event was defined as any untoward medical occurrence in a participant, temporally associated with the use of an investigational product, whether or not considered related to the investigational product.
Time Frame: For 140.57 weeks at maximum, starting from Week 24
Population: Safety Population: Participants who had received at least one dose of the investigational product
Measure: Number; unit: participants
Arm/Group | GSK1325760A
Number analyzed (Participants) | 21
participants | 21

2. Secondary Outcome: Mean Change From Baseline in Six Minutes Walk Distance (6MWD) at Weeks 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, and 156
Description: Change from baseline was calculated as each value at Weeks 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, and 156 minus the baseline value. 6MWD was measured by a 6-minute walk test. This test measures the distance that a participant can walk in a period of 6 minutes. Imputation technique was last observation carried forward, which was used in an attempt to compensate for missing data. For each participant, missing values were replaced with the last observed value.
Time Frame: Baseline and Weeks 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, and 156
Population: Full Analysis Set (FAS): All participants registered, with the exception of those who did not receive any dose of the investigational product and those who had no efficacy assessment after treatment.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | GSK1325760A
Number analyzed (Participants) | 21
meters
  Week 24 | 53.55 (52.951)
  Week 36 | 51.90 (61.141)
  Week 48 | 59.61 (53.415)
  Week 60 | 46.38 (56.871)
  Week 72 | 59.86 (59.667)
  Week 84 | 58.11 (64.244)
  Week 96 | 49.84 (57.571)
  Week 108 | 56.38 (67.131)
  Week 120 | 58.66 (66.633)
  Week 132 | 54.42 (66.402)
  Week 144 | 54.83 (67.739)
  Week 156 | 49.19 (78.369)

3. Secondary Outcome: Mean Change From Baseline in the Borg Dyspnea Index (BDI) at Weeks 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156, and Withdrawal/Completion
Description: The BDI was calculated by using a 10-point scale (0 = None, 10 = Maximum) and indicates the degree of breathlessness after completion of the 6-minute walk test. The BDI scale was assessed by each participant. Change from baseline was calculated as each value at Weeks 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156, and Withdrawal/Completion minus the baseline value. Observed data analysis (no imputation technique).
Time Frame: Baseline and Weeks 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156, and Withdrawal/Completion (up to Week 159.85)
Population: FAS. Participants were followed for different lengths of time; thus, not all participants were analyzed at all study weeks.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | GSK1325760A
Number analyzed (Participants) | 21
scores on a scale
  Week 24, n=21 | -0.79 (1.670)
  Week 36, n=21 | -0.57 (2.254)
  Week 48, n=20 | -1.00 (2.242)
  Week 60, n=21 | -1.00 (2.372)
  Week 72, n=18 | -1.08 (2.433)
  Week 84, n=18 | -1.31 (2.438)
  Week 96, n=17 | -0.74 (2.617)
  Week 108, n=18 | -0.58 (2.574)
  Week 120, n=16 | -0.94 (2.732)
  Week 132, n=10 | 1.30 (2.371)
  Week 144, n=7 | 1.21 (1.776)
  Week 156, n=4 | -0.13 (1.436)
  Withdrawal/Completion, n=7 | -0.36 (4.308)

4. Secondary Outcome: Number of Participants With the Indicated Change From Baseline in Their World Health Organization (WHO) Functional Classification (FC) at Weeks 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156, and Withdrawal/Completion
Description: There are four grades for the WHO FC (Class I = none, Class IV = most severe). The WHO FC indicates the severity of Pulmonary Arterial Hypertension and is an adaptation of the New York Heart Association classification. It was assessed by the investigator. Observed data analysis (no imputation technique).
Time Frame: Baseline and Weeks 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156, and Withdrawal/Completion (up to Week 164.14)
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | GSK1325760A
Number analyzed (Participants) | 21
participants
  Improved at Week 24, n=21 | 10
  No change at Week 24, n=21 | 11
  Deteriorated at Week 24, n=21 | 0
  Improved at Week 36, n=21 | 10
  No change at Week 36, n=21 | 11
  Deteriorated at Week 36, n=21 | 0
  Improved at Week 48, n=21 | 11
  No change at Week 48, n=21 | 9
  Deteriorated at Week 48, n=21 | 1
  Improved at Week 60, n=21 | 11
  No change at Week 60, n=21 | 10
  Deteriorated at Week 60, n=21 | 0
  Improved at Week 72, n=20 | 8
  No change at Week 72, n=20 | 12
  Deteriorated at Week 72, n=20 | 0
  Improved at Week 84, n=19 | 9
  No change at Week 84, n=19 | 10
  Deteriorated at Week 84, n=19 | 0
  Improved at Week 96, n=19 | 9
  No change at Week 96, n=19 | 10
  Deteriorated at Week 96, n=19 | 0
  Improved at Week 108, n=19 | 9
  No change at Week 108, n=19 | 10
  Deteriorated at Week 108, n=19 | 0
  Improved at Week 120, n=18 | 8
  No change at Week 120, n=18 | 10
  Deteriorated at Week 120, n=18 | 0
  Improved at Week 132, n=13 | 5
  No change at Week 132, n=13 | 8
  Deteriorated at Week 132, n=13 | 0
  Improved at Week 144, n=10 | 3
  No change at Week 144, n=10 | 7
  Deteriorated at Week 144, n=10 | 0
  Improved at Week 156, n=6 | 2
  No change at Week 156, n=6 | 4
  Deteriorated at Week 156, n=6 | 0
  Improved at Withdrawal/Completion, n=20 | 10
  No change at Withdrawal/Completion, n=20 | 10
  Deteriorated at Withdrawal/Completion, n=20 | 0

5. Secondary Outcome: Number of Participants With the Indicated Event, as an Assessment of Time to Clinical Worsening of Pulmonary Arterial Hypertension (PAH), Assessed as the First Occurrence of a Particular Event
Description: Time to clinical worsening was defined as the time from baseline to the first occurrence of death, lung transplantation, hospitalization for PAH treatment, atrial septostomy (a surgical procedure in which a small hole is made in the wall between the left and right atria of the heart), or study discontinuation due to change to other PAH treatment. Time to clinical worsening was measured as the number of participants who experienced these events up to 164.14 weeks.
Time Frame: Up to 164.14 weeks
Population: FAS
Measure: Number; unit: participants
Arm/Group | GSK1325760A
Number analyzed (Participants) | 21
participants
  Death | 0
  Lung transplantation | 0
  Hospitalization for PAH treatment | 0
  Atrial septostomy | 0
  Study discontinuation (additional medication) | 1

6. Secondary Outcome: Mean Change From Baseline in Mean Pulmonary Artery Pressure (mPAP) at Weeks 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156, and Withdrawal/Completion
Description: mPAP is a measure of cardiopulmonary hemodynamics (echocardiography). Change from baseline was calculated as each value at Weeks 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156, and Withdrawal/Completion minus the baseline value. Observed data analysis (no imputation technique).
Time Frame: Baseline and Weeks 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156, and Withdrawal/Completion (up to Week 153)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | GSK1325760A
Number analyzed (Participants) | 19
millimeters of mercury (mmHg)
  Week 24, n=19 | -9.96 (7.419)
  Week 36, n=19 | -8.16 (8.969)
  Week 48, n=19 | -7.06 (10.064)
  Week 60, n=18 | -5.44 (14.839)
  Week 72, n=18 | -10.68 (10.661)
  Week 84, n=15 | -9.23 (14.241)
  Week 96, n=16 | -13.33 (13.108)
  Week 108, n=16 | -10.87 (10.786)
  Week 120, n=15 | -10.56 (10.011)
  Week 132, n=10 | -13.30 (10.592)
  Week 144, n=8 | -12.04 (9.364)
  Week 156, n=6 | -13.85 (8.900)
  Withdrawal/Completion, n=6 | -10.72 (14.972)

7. Secondary Outcome: Mean Change From Baseline in Cardiac Output (CO) at Weeks 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156, and Withdrawal/Completion
Description: CO is a measure of cardiopulmonary hemodynamics (echocardiography). Change from baseline was calculated as each value at Weeks 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156, and Withdrawal/Completion minus the baseline value. Observed data analysis (no imputation technique).
Time Frame: Baseline and Weeks 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156, and Withdrawal/Completion (up to Week 156.14)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Liters per minute (L/min)
Arm/Group | GSK1325760A
Number analyzed (Participants) | 20
Liters per minute (L/min)
  Week 24, n=20 | 0.425 (1.6453)
  Week 36, n=20 | 0.291 (1.6786)
  Week 48, n=20 | 0.227 (1.5546)
  Week 60, n=20 | 0.430 (1.2865)
  Week 72, n=19 | -0.002 (1.4237)
  Week 84, n=18 | 0.151 (1.5211)
  Week 96, n=18 | 0.025 (1.3813)
  Week 108, n=17 | 0.175 (1.6398)
  Week 120, n=17 | 0.285 (1.2126)
  Week 132, n=13 | 0.068 (1.4774)
  Week 144, n=10 | 0.391 (1.1643)
  Week 156, n=5 | 0.458 (0.5779)
  Withdrawal/Completion, n=7 | 0.257 (1.1571)

8. Secondary Outcome: Mean Change From Baseline in B-type Natriuretic Peptide (BNP) Values at Weeks 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156, and Withdrawal/Completion
Description: Change from baseline was calculated as each value at Weeks 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156, and Withdrawal/Completion minus the baseline value. BNP is a surrogate marker of heart failure and was measured by a central laboratory. Observed data analysis (no imputation techniques).
Time Frame: Baseline and Weeks 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156, and Withdrawal/Completion (up to Week 164.14)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: nanograms per liter (ng/L)
Arm/Group | GSK1325760A
Number analyzed (Participants) | 21
nanograms per liter (ng/L)
  Week 24, n=20 | -109.54 (170.495)
  Week 36, n=21 | -96.98 (167.736)
  Week 48, n=21 | -70.40 (211.457)
  Week 60, n=21 | -79.89 (232.876)
  Week 72, n=20 | -81.36 (204.379)
  Week 84, n=19 | -118.78 (160.738)
  Week 96, n=19 | -115.73 (146.038)
  Week 108, n=19 | -117.07 (183.770)
  Week 120, n=18 | -113.23 (164.368)
  Week 132, n=13 | -140.93 (215.436)
  Week 144, n=10 | -138.17 (226.688)
  Week 156, n=6 | -146.52 (218.553)
  Withdrawal/Completion, n=20 | -62.72 (260.373)

9. Primary Outcome: Number of Participants With Adverse Events Categorized by Severity
Description: The severity of adverse events was assessed by the investigator; events were assigned to one of the following categories: mild, an event that was easily tolerated by the participant, causing minimal discomfort and not interfering with everyday activities; moderate, an event that was sufficiently discomforting to interfere with normal everyday activities; and severe, an event that prevented normal everyday activities.
Time Frame: For 140.57 weeks at maximum, starting from Week 24
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | GSK1325760A
Number analyzed (Participants) | 21
participants
  Mild | 12
  Moderate | 5
  Severe | 4

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs were collected for 140.57 weeks at maximum, starting from Week 24.
Arm/Group | GSK1325760A
Serious Adverse Events (participants affected / at risk) | 8/21
Other Adverse Events (participants affected / at risk) | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GSK1325760A (N=21)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Ventricular tachycardia (Cardiac disorders) | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1
Sudden hearing loss (Ear and labyrinth disorders) | 1
Vitreous haemorrhage (Eye disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hepatic encephalopathy (Nervous system disorders) | 1
Renal failure (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GSK1325760A (N=21)
Nasopharyngitis (Infections and infestations) | 18
Pyrexia (General disorders) | 8
Back pain (Musculoskeletal and connective tissue disorders) | 7
Diarrhoea (Gastrointestinal disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Gastroenteritis (Gastrointestinal disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Dizziness (Nervous system disorders) | 3
Headache (Nervous system disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 3
Cystitis (Infections and infestations) | 2
Onychomycosis (Infections and infestations) | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Abdominal discomfort (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Toothache (Gastrointestinal disorders) | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 2
Eczema (Skin and subcutaneous tissue disorders) | 2
Anaemia (Blood and lymphatic system disorders) | 2
Leukopenia (Blood and lymphatic system disorders) | 2
Flushing (Vascular disorders) | 2
Hot flush (Vascular disorders) | 2
Vertigo (Ear and labyrinth disorders) | 2
Hepatic function abnormal (Hepatobiliary disorders) | 2
Joint sprain (Injury, poisoning and procedural complications) | 2
Decreased appetite (Metabolism and nutrition disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.